CLINICAL TRIAL: NCT00317460
Title: On-Site Addiction Treatment With Buprenorphine in HIV Clinical Care Settings
Brief Title: Buprenorphine and Integrated HIV Care
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: The New York Academy of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0510000681
Record Dates: First submitted 2006-04-20; First posted 2006-04-24 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Substance-related Disorders; Drug Addiction; Human Immunodeficiency Virus; AIDS; HIV Infections
Keywords: Drug Abuse; Drug Addiction; Drug Dependence; Drug Use Disorders; Drug Use Disorder; Substance Abuse; Substance Use Disorder; Buprenorphine; Opiate Addiction
MeSH Terms: conditions — Substance-Related Disorders; Acquired Immunodeficiency Syndrome; HIV Infections; Opioid-Related Disorders | interventions — Practice Management; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Physician Management
  Interventions: Other: Physician Management
- 2 (Experimental): Physician Management and counseling (drug counseling and medication adherence)
  Interventions: Behavioral: Counseling

INTERVENTIONS:
Other: Physician Management — Standard physician care
  Arms: 1
Behavioral: Counseling — Physician Management and Counseling
  Arms: 2

SUMMARY:
The purpose of this study is to examine the efficacy of providing two levels of psychosocial support along with buprenorphine/naloxone (BUP) maintenance to opioid dependent patients receiving their care in an HIV clinical care setting.

DETAILED DESCRIPTION:
The purpose of this study is to examine the efficacy of providing two levels of psychosocial support along with buprenorphine/naloxone (BUP) maintenance to opioid dependent patients receiving their care in an HIV clinical care setting. The proposed study will compare Physician Management (PM), a manual-guided brief intervention that approximates the usual counseling provided by primary care practitioners to patients with chronic medical conditions vs. an enhanced strategy of PM with the addition of a combined drug counseling and adherence management strategy (PM+DC/AM). DC is designed to educate the patient about the recovery process and provide additional advice about lifestyle changes including HIV transmission risk reduction and 12-step participation. Adherence Management (AM) is a counseling strategy focusing on HIV medication adherence, adapted from Sorensen et al1. This research will build on pilot work that is being completed in order to further develop and refine these counseling interventions, determine what other psychosocial interventions might be required, and to evaluate this model of integrated care in terms of its effects on opioid agonist therapy retention, decreasing illicit drug use, and increasing adherence to highly active antiretroviral therapy (HAART). Finally, it will provide data that will aid in the formulation of guidelines and the creation of practical manuals for optimizing the provision of this novel therapy to individuals with HIV disease and opioid dependence, as well as provide data for future funded randomized clinical trials.

From September 2005 (start date) to December 1, 2007, the study was conducted as part of a multi-site project that was overseen by the New York Academy of Medicine (NYAM), which is in charge of data analysis. Following December 1, 2007, the study will continue as a local, single-site project without further collaboration from NYAM.

ELIGIBILITY:
Inclusion Criteria:

* HIV disease
* DSM-IV criteria for opioid dependence, as assessed by SCID
* Documented opioid positive urine toxicology testing

Exclusion criteria:

* Desire to remain enrolled in opioid agonist treatment at an opioid treatment program
* Current dependence on alcohol, benzodiazepines or sedatives (patients who are receiving benzodiazepines under the care of a psychiatrist for the treatment of an anxiety disorder will not be excluded)
* Current suicide or homicide risk
* Current psychotic disorder or major depression
* Inability to read or understand English
* Dementia
* Life-threatening or unstable medical problems requiring inpatient medical care or nursing home placement
* Currently enrolled in other studies involving the provision of psychosocial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2005-09; Primary Completion 2009-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Treatment retention | 52 weeks
Reductions in illicit opioid use | 52 weeks
Adherence to antiretroviral medications | 52 weeks

SECONDARY OUTCOMES:
T-lymphocyte CD4 cell count | 52 weeks
HIV-1 RNA levels | 52 weeks
Reduction in HIV transmission risk behaviors | 52 weeks
Improved health status | 52 weeks
Patient satisfaction | 52 weeks
Provider satisfaction | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Cutter, Ph.D., Study Director — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- See also: Click here for more information about this study: Buprenorphine and Integrated HIV Care Evaluation and Support Center (BHIVES). — http://www.bhives.org